CLINICAL TRIAL: NCT07281001
Title: A Study to Assess the Efficiency of Trastuzumab Deruxtecan in Russian Breast Cancer Patients
Acronym: Traderrus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 29.11.2025
Record Dates: First submitted 2025-11-29; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: HER2-positive Breast Cancer; Trastuzumab Deruxtecan
Keywords: Trastuzumab Deruxtecan; HER2-positive Breast Cancer
MeSH Terms: interventions — Isovaleryl-CoA Dehydrogenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with unresectable or metastatic HER2+ BC who have received one or more cycles T-DXd (Experimental)
  Interventions: Drug: T-DXd 5.4 mg/kg, IVD, 1 cycle every 21 days.

INTERVENTIONS:
Drug: T-DXd 5.4 mg/kg, IVD, 1 cycle every 21 days. — T-DXd 5.4 mg/kg, IVD, 1 cycle every 21 days. Intravenous infusion

SUMMARY:
This multi-center observational retrospective study will collect real-world clinical data from eligible patients with unresectable or metastatic HER2+ breast cancer who have received one or more cycles Trastuzumab Deruxtecan in Russian Federation

DETAILED DESCRIPTION:
This multi-center observational retrospective study will collect real-world clinical data from eligible patients with unresectable or metastatic HER2+ breast cancer who have received one or more cycles Trastuzumab Deruxtecan in Russian Federation

The aim of this trial is to explore the real-world effectiveness T-Dxd and potential predictors in Russian metastatic breast cancer patients

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged over 18 years old.
2. Metastatic breast cancer included unresectable locally advanced breast cancer, de novo stage IV breast cancer, and recurrent metastatic breast cancer.
3. Patients has received Trastuzumab Deruxtecan
4. Available medical history.

Exclusion Criteria:

1. Incomplete medical history.
2. Pregnancy or breast-breeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
PFS | 6 weeks
  progression-free survival

SECONDARY OUTCOMES:
ORR | 6 weeks
  Overall Response Rate
CBR | 6 weeks
  Clinical benefit Rates
OS | 6 weeks
  Overall Survival
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 weeks
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Elena Artamonova, Principal Investigator — The Blokhin National Medical Research Center of Oncology of the Russian Ministry of Health
Locations (1):
- Federal State Budgetary Institution "N.N. Blokhin National Medical Research Center of Oncology" оf the Ministry of Health of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No